CLINICAL TRIAL: NCT01267591
Title: Peripheral Artery Tonometry in Children With Type 1 Diabetes and Obese Children.
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: kristina casteels, Pediatrie, UZLeuven
Other Study IDs: UZLeuven
Record Dates: First submitted 2010-12-27; First posted 2010-12-28 (Estimated); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Peripheral Artery Tonometry; Diabetes; Children; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- control
- type 1 diabetes
- obesity

SUMMARY:
Background: The reactive hyperemia-peripheral artery tonometry (RH-PAT) is a newly developed method for noninvasive endothelial function assessment.

Objective: The goal of this study is to determine whether a significant difference in RH-PAT score is present between adolescents with type 1 diabetes (T1D) in comparison with controls. We will also compare RH-PAT scores in obese adolescents versus controls.

ELIGIBILITY:
Inclusion Criteria:

* 12-19 years of age

Exclusion Criteria:

* type 2 diabetes; obesity in group of type 1 diabetes

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children seen at consultation in University Hospital
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2009-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
RHPAT | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Pareyn A, Allegaert K, Verhamme P, Vinckx J, Casteels K. Impaired endothelial function in adolescents with overweight or obesity measured by peripheral artery tonometry. Pediatr Diabetes. 2015 Mar;16(2):98-103. doi: 10.1111/pedi.12139. Epub 2014 Apr 3. PMID 24698176